CLINICAL TRIAL: NCT02524379
Title: Spinal Cord Injury Neuroprotection With Glyburide; Pilot Study: An Open-Label Prospective Evaluation of the Feasibility, Safety, Pharmacokinetics, and Preliminary Efficacy of Oral Glyburide (DiaBeta) in Patients With Acute Traumatic Spinal Cord Injury
Brief Title: Spinal Cord Injury Neuroprotection With Glyburide
Acronym: SCING
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Principal investigator has left the university; there were not enough participants to analyze the data.
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014H0335
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Acute Spinal Cord Injury
MeSH Terms: interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glyburide Treatment Arm (Experimental): Enrolled patients will receive 12 doses of Glyburide starting within 8 hours of SCI. The dosing regimen involves an initial dose of 1.25 mg followed by eleven consecutive doses of 0.625 mg every 6 hours. The total daily dose of Glyburide on Day 1, Day 2 and Day 3 will be 3.125 mg, 2.5 mg, and 2.5 mg respectively.
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: Glyburide — 3 day drug regimen beginning 8 hours after acute traumatic spinal cord injury.

SUMMARY:
The purpose of this study is to determine the safety of using oral Glyburide in patients with acute traumatic cervical spinal cord injuries (SCI).

DETAILED DESCRIPTION:
This study will include patients between 18 and 80 years who have experienced acute traumatic cervical spinal cord injury (specifically ASIA A, B or C). Patients will then begin an oral drug regimen of Glyburide, which must be started within 8 hours of injury and continued for 72 hours at a daily dose of 3.125 mg on Day 1, 2.5 mg on Day 2 and 2.5 mg on Day 3. If indicated, the patient will also have surgical intervention for spinal cord decompression and spinal stabilization. Each patient who takes part in this study will have labs drawn regularly and adverse events assessed daily through Day 14 or discharge (whichever is earlier). Study participation will last for 365 days (+/- 30 days), with post-hospitalization follow-up occurring on Days 28, 42, 84, 182 and 365.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years and ≤ 80 years
2. Written informed consent by patient or legal authorized representative
3. No other life-threatening injury
4. No evidence of sepsis
5. Acute cervical SCI with ASIA Impairment Scale grade A, B or C on admission
6. Non-penetrating SCI at neurologic level from C2 to C8
7. Initiation of study drug within 8 hours of injury

Exclusion Criteria

1. Unconsciousness or other mental impairment that prevents neurological assessment within the first 8 hours
2. Acute SCI with ASIA Impairment Scale grade D or E
3. Currently involved in another non-observational SCI research study or receiving another investigational drug
4. History of hypersensitivity to sulfonylureas, in particular glyburide, or any of its components
5. Other illness (including mental disorder) that could preclude accurate medical and neurological evaluation (at discretion of the site investigator)
6. Unable to commit to the follow-up schedule
7. A recent history of regular substance abuse (illicit drugs, alcohol), which in the opinion of the investigator would interfere with the subject's participation in the study
8. Any condition likely to result in the patient's death within the next 12 months
9. Prisoner
10. Severe renal disorder from the patient's history (e.g. dialysis) or baseline eGFR of < 30 mL/min/1.73 m2
11. Known severe liver disease, or ALT > 3 times upper limit of normal or bilirubin > 2 times upper limit normal. Subjects may be randomized if liver function tests have been drawn but are not yet available and the subject has no known history of liver disease; however, treatment with DiaBeta will be discontinued prior to the second dose if liver function tests indicate ALT > 3 times upper limit of normal or bilirubin > 2 times upper limit of normal
12. Blood glucose <55 mg/dL at enrollment or immediately prior to administration of DiaBeta, or a clinically significant history of hypoglycemia
13. Acute ST elevation myocardial infarction, and/or acute decompensated heart failure, and/or QTc > 520 ms, and/or known history of cardiac arrest (PEA, VT, VF, asystole), and/or admission for an acute coronary syndrome, myocardial infarction, or coronary intervention (percutaneous coronary intervention or coronary artery surgery) within the past 3 months
14. Known treatment with Bosentan within past 7 days
15. Known G6PD enzyme deficiency
16. Pregnancy: Women must be either post-menopausal, permanently sterilized or, if ≤ 50 years old, must have a negative test for pregnancy obtained before enrollment
17. Breast-feeding women who do not agree to stop breast-feeding during and for 7 days following the end of oral glyburide administration
18. Subjects who in the opinion of the investigator are not suitable for inclusion in the study (reason to be documented).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Francis Farhadi, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Minnema AJ, Mehta A, Boling WW, Schwab J, Simard JM, Farhadi HF. SCING-Spinal Cord Injury Neuroprotection with Glyburide: a pilot, open-label, multicentre, prospective evaluation of oral glyburide in patients with acute traumatic spinal cord injury in the USA. BMJ Open. 2019 Oct 10;9(10):e031329. doi: 10.1136/bmjopen-2019-031329. PMID 31601596

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glyburide Treatment Arm
Started | 3
Completed | 2
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glyburide Treatment Arm
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With tSCI Recruited Within the Specified Time Window
Description: A measure of feasibility of undertaking a larger phase II study among this population of patients where treatment must begin within a short injury-to-drug time window.
Time Frame: Enrollment Period (within 8 hours of tSCI)
Population: A total of 24 patients with acute cervical tSCI were screened over the course of the study for eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Glyburide Treatment Arm
Number analyzed (Participants) | 24
Participants | 3

2. Primary Outcome: Number of Drug Related Adverse Events
Description: A measure of safety of treating patients with traumatic spinal cord injury with Glyburide administered orally within a short injury-to-drug time window.
Time Frame: One year post enrollment
Measure: Number; unit: Events
Arm/Group | Glyburide Treatment Arm
Number analyzed (Participants) | 3
Events | 0

3. Secondary Outcome: Number of Participants With Neurologic Recovery Following tSCI
Description: The neurologic status of patients will be assessed using the American Spinal Injury Association (ASIA) Impairment Scale (AIS) as assessed by International Standards for Neurological Classification of SCI (ISNCSCI) criteria.
Time Frame: One year post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Glyburide Treatment Arm
Number analyzed (Participants) | 2
Participants | 2

4. Secondary Outcome: Serum Pharmacokinetic and Biomarker Analysis
Description: Plasma concentrations will be serially quantified through day 3 following tSCI to evaluate the pharmacokinetics of Glyburide in the acute tSCI population. Comparisons will be made to reported levels achieved in healthy patient cohorts. Standard enzyme-linked immunosorbent assay (ELISA) techniques will be used to measure blood levels of neurofilament light chain, neuron- specific enolase, tau, S100b, and glial fibrillary acidic protein levels on admission, at 24 hours and on days 3 and 7 following tSCI to evaluate serum biomarker levels. Comparisons will be made to previously published values observed in non-treated control patients
Time Frame: Enrollment through post-treatment day 7
Population: Principal Investigator left university: Samples were not analyzed at study termination.
Arm/Group | Glyburide Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Glyburide Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glyburide Treatment Arm (N=3)
Bradycardia (Cardiac disorders) | 1 (1)
Other Dysrhythmia (Tachy-brady syndrome) (Cardiac disorders) | 1 (1)
Acute Renal Failure (Gastrointestinal disorders) | 1 (1)
Acute respiratory distress syndrome (ARDS) - Atelecetasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glyburide Treatment Arm (N=3)
Thromocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Urinary Tract Infection (UTI) (Infections and infestations) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT02524379/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT02524379/ICF_001.pdf